CLINICAL TRIAL: NCT02120989
Title: A Pilot Study Examining the Effectiveness of Partner-Assisted Cognitive Behavioral Therapy for Insomnia
Brief Title: Researching Effective Sleep Treatments (Project REST)
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Veterans Medical Research Foundation (Other); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sean P.A. Drummond, Associate Professor of Psychiatry, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H140059
Record Dates: First submitted 2014-04-11; First posted 2014-04-23 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia
Keywords: insomnia; cognitive behavioral therapy for insomnia (CBT-I); partner-assisted
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Partner-Assisted Cognitive Behavioral Therapy for Insomnia — Study treatment includes partner-assisted Cognitive Behavioral Therapy for Insomnia (CBT-I) and consists of 7-8 weekly group therapy sessions of 2 hours each. Partner-assisted CBT-I focuses on altering patients' sleep schedules and changing their behaviors and patterns around sleeping in order to help them sleep in a single block of time overnight. As part of this treatment, participants will be asked to change, possibly reduce, the amount of time spent in bed and to maintain a specific bed time and wake time, as well as other potential changes depending on his/her specific insomnia pattern. This treatment has been shown to be safe and efficacious for a wide range of patients.

SUMMARY:
We will undertake initial development of a new behavioral sleep intervention (i.e., partner-assisted Cognitive Behavioral Therapy for Insomnia; CBT-I), based closely on the gold standard treatment, CBT-I. We will examine if the new treatment has a positive impact on subjective and objective sleep and quality of life in a clinic-based sample. Secondary aims will examine treatment adherence and maintenance of therapeutic gains as well as relationship satisfaction and broader psychiatric functioning.

DETAILED DESCRIPTION:
Objective: To investigate whether partner-assisted Cognitive Behavioral Therapy for Insomnia (CBT-I) has a positive impact on subjective and objective sleep and quality of life in individuals with insomnia. Secondary aims will examine treatment adherence and maintenance of therapeutic gains as well as relationship satisfaction and impact on broader psychiatric functioning.

Research Design: This is an open trial, feasibility study designed to examine the effectiveness of partner-assisted CBT-I on insomnia patient's sleep and quality of life. After individuals, Veterans and non-Veterans, and their respective bed partners consent to participate in this treatment study, we will collect de-identified data including self-report questionnaires, daily sleep diaries, and actigraphy (ambulatory sleep/wake monitoring). For Veteran participants, we also plan to collect data from medical records. Study participants will be seen for study partner-assisted CBT-I treatment at the VA San Diego Healthcare System (VASDHS) Sleep and Mood Clinic. The initial screening appointment and 1-month follow up assessment will be conducted in the Veterans Medical Research Foundation (VMRF) building. The entire study will take two years; participation for Veterans and non-Veterans will last about 3 months from the date of initial screening appointment to their follow up assessment.

Methodology:

Procedures:

Participants will primarily be recruited through the VASDHS's Sleep and Mood Clinic by physician and clinician referrals as well as posted study fliers in these clinics. Non-veterans such as those enrolled in other UCSD research studies will also be recruited. All individuals who meet eligibility criteria will be offered the opportunity to participate and informed consent will be obtained for those who wish to do so. Participation or non-participation in the protocol will not affect clinical care. Assessments of sleep symptoms, health-related quality of life, treatment adherence, relationship satisfaction, and psychiatric functioning will occur as part of standard treatment protocols. Assessments include self-report questionnaires as well as weekly sleep diaries and two weeks of actigraphy (e.g., at the start and end of treatment). Assessment data will be de-identified and analyzed to determine: (a) descriptive characteristics of study participants; (b) effectiveness of partner-assisted CBT-I treatment; (c) relationship functioning; (d) treatment adherence (e.g., did participants follow treatment recommendations from week to week); and, (e) any reduction in symptoms of psychiatric conditions that frequently co-occur with insomnia including mood and/or PTSD symptoms.

Treatment:

We aim to test the effectiveness of partner-assisted CBT-I treatment in patients with insomnia. There are currently no published studies on a couple-based CBT-I approach. The proposed treatment will closely resemble the CBT-I manual currently used for insomnia group therapy in the VA Sleep and Mood Clinic. The main difference will be the inclusion of patients' partners in treatment and administering the manual with emphasis on how patients' partners can assist the patient in making behavioral changes outlined and prioritized in the existing manual.

Data Extraction and Security Plan:

Data will be collected and extracted in a de-identified format and coded only with a study specific number.

* Demographic information: e.g., age, relationship status, era of military service (for Veteran participants), gender, race and ethnicity.
* Treatment information: e.g., number of sessions attended, treatment adherence, treatment barriers.
* Medical / Psychiatric Information: e.g., history of treatment for psychiatric co-morbidities, use of pharmacological agents, and presence of medical conditions.

Statistical Procedures:

* Prior to quantitative analyses, data will be screened to ensure quality and to check standard statistical assumptions.
* Descriptive Statistics will be used to calculate frequency of demographic variables in patients.
* Paired sample t-tests will examine change in pre-treatment and post-treatment means for sleep, quality of life and relationship satisfaction variables.
* Paired sample t-tests will also examine change in post-treatment and follow-up means for sleep, quality of life and relationship satisfaction variables.
* Descriptive Statistics will calculate average weekly treatment adherence from the participant, partner and the therapist perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Meet diagnostic criteria for insomnia, including a score of 8 or higher on the Insomnia Severity Index (ISI)
* Stable bed partner (i.e., someone with whom they have lived for at least one month prior to the screening appointment and someone who they anticipate to continue living with for the next two months while in the study treatment) who can commit to participating in patient's insomnia treatment. Patients and bed partners who sleep in different beds are eligible to participate.
* English literacy
* Participation in the group Partner-Assisted Cognitive Behavioral Therapy for Insomnia (CBT-I) class

Exclusion Criteria:

* A score of 7 or lower on the Insomnia Severity Index (ISI)
* Unmanaged psychosis or manic episodes in the past two months. For any interested potential participants with a history of bipolar disorder, their bipolar disorder must be stable (i.e., euthymic) for two months in order to be eligible to participate.
* Diagnosed (previously or by our study screen) and untreated sleep disorder other than insomnia. Sleep disorders diagnosed, but stably treated (e.g., obstructive sleep apnea treated with CPAP) will be allowed, as long as the treatment is not a hypnotic medication.
* Severe medical or psychiatric illness that would make it difficult to regularly attend psychotherapy sessions or participate fully in the study
* Current substance use disorder, or meeting criteria for a SUD within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Functioning from Baseline to the End of Treatment | baseline; treatment week 4; week 8 (at end of treatment); 1 month post-treatment follow-up
  Primary outcome measures (see below for more information about the measures) will assess the change in sleep functioning from baseline to the end of treatment. We will also examine change in sleep functioning from baseline to the 1-month post treatment assessment.
  Sleep diaries. Participants will be asked to complete a daily sleep diary throughout the 8 week treatment and one week prior to the 1 month post-treatment follow up appointment. Each morning participants are asked to record sleep habits, such as bedtime, wake time, time in bed, and number and duration of awakenings. Our sleep diary will include questions to track treatment adherence. Sleep diaries are widely used in studies of insomnia.
  Questionnaire. Insomnia Severity Index (ISI; Morin et al., 2011). The ISI consists of 7-items that assess severity of insomnia, satisfaction with sleep pattern, effect of sleep on daytime and social functioning, and concern about current sleep difficulties in the past week.

SECONDARY OUTCOMES:
Change in Quality of Life from Baseline to the End of Treatment | baseline; treatment week 4; week 8 (at end of treatment); 1 month post-treatment follow-up
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF; Endicott, Nee, Harrison, & Blumentha, 1993). The Q-LES-Q-SF is a 16-item self-report questionnaire assessing quality of life on multiple domains over the past week including physical and mental health as well as satisfaction with relationships, activities, and overall sense of well being. It has demonstrated good validity.
Change in Relationship Functioning from Baseline to the End of Treatment | baseline; treatment week 4; week 8 (at end of treatment); 1 month post-treatment follow-up
  Dyadic Adjustment Scale (DAS; Spanier, 1976). The DAS is a 32-item inventory of relationship adjustment in couples. It is a widely used measure with sound psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Sean PA Drummond, PhD, Principal Investigator — VA San Diego Healthcare System and University of California San Diego; Melissa M Jenkins, PhD, Study Director — VA San Diego Healthcare System and University of California San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] Smith MT, Perlis ML, Park A, Smith MS, Pennington J, Giles DE, Buysse DJ. Comparative meta-analysis of pharmacotherapy and behavior therapy for persistent insomnia. Am J Psychiatry. 2002 Jan;159(1):5-11. doi: 10.1176/appi.ajp.159.1.5. PMID 11772681
- [Background] Perlis, M.L., et al., Cognitive-behavioral therapy for insomnia, in Clinical Handbook of Insomnia. 2004, Springer. p. 155-171.
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Spanier, G.B., Measuring Dyadic Adjustment: New Scales for Assessing the Quality of Marriage and Similar Dyads. Journal of Marriage and Family, 1976. 38(1): p. 15-28.